CLINICAL TRIAL: NCT02119481
Title: Effects of Mindfulness Meditation and Stress Management Training on Perceived Stress, Psychological Well-being, and Sleep Quality Among Patients Diagnosed With Breast Cancer
Brief Title: Effects of Mindfulness Meditation and Stress Management After Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Richard Branstrom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KI-MBSR-Main-BC
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: Mindfulness stress reduction training; Expressive writing condition; Waiting list control condition
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness-based stress reduction (Experimental): Mindfulness-based stress reduction training
  Interventions: Behavioral: Mindfulness-based stress reduction
- Expressive writing condition (Active Comparator): Expressive writing
  Interventions: Behavioral: Expressive writing condition
- Waiting-list control condition (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction
  Other Names: MBSR; MBCT; Mindfulness based cognitive behavioral therapy
  Arms: Mindfulness-based stress reduction
Behavioral: Expressive writing condition
  Other Names: Expressive writing
  Arms: Expressive writing condition

SUMMARY:
The primary aim of this study is to examine the effects of a mindfulness-based stress reduction training program, delivered in individual web-based sessions, among breast cancer patients. The objectives are to study and answer questions regarding effects of the such training in a randomized controlled trial including the following outcome measures: physical and mental health status, perceived stress, post-traumatic stress symptoms, psychological well-being, and sleep quality. In addition to the primary aim, the investigators plan to explore potential mechanisms through which mindfulness training lead to improvement in perceived stress, well-being and sleep-quality. This will be studied by mediational analyses.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient ≥ 18 years of age who has received the cancer diagnosis ≤ 2 years previously
* Access and regular use of the internet

Exclusion Criteria:

* Non Swedish speaking
* Previous sever psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-05; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress | Baseline to 8 week follow-up change
  Perceived stress as measured with the Perceived stress scale (PSS) and the Intrusion of event scale revised (IES-R) before and after intervention
Change in Psychological Well-Being | Baseline to 8 week follow-up change
  Psychological Well-Being as measured with the Psychological Well-Being (PWB) scale by C Ryff; a questionnaire measuring six dimensions of psychological well-being: environmental mastery; self-acceptance; positive relations with others; purpose in life; personal growth; and autonomy.
Change in Sleep quality | Baseline to 8 week follow-up change
  Sleep quality as measured with the Karolinska Sleep Questionnaire (KSQ) a 13-item questionnaire assessing sleep-time and quality as well as perceived satisfaction with sleep, sleepiness and sleep disturbance.

SECONDARY OUTCOMES:
Change in Perceived stress | Change from baseline to 12 months follow-up
  Change in Perceived stress as measured with the Perceived stress scale and the Intrusion of event scale revised (IES-R)
Change in Psychological well-being | Change from baseline to 12-month follow-up
  Change in psychological well-being as measured with the Psychological well-being scale.
Change in Sleep quality | Change from baseline to 12-month follow-up
  Change in sleep quality as measured with the Karolinska sleep questionnaire.

OTHER OUTCOMES:
Sickness-absence for work | At 24 months follow-up
  Gorup differences in sickness-absence from work as measured in national population registries
All cause morbidity | At 24 months follow-up
  Group differences in all cause morbidity as measured in national registries
All cause mortality | At 24 months follow-up
  Group differences in all cause mortality as measured in national registries.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Department of clinical neuroscience, Stockholm, Sweden